CLINICAL TRIAL: NCT01244620
Title: A Phase 1, Open Label, Randomized, Four Period, Crossover, Multiple Dose Study To Assess The Pharmacokinetic Interaction Between Sitaxsentan and Tadalafil and The Effect Of Sildenafil On Sitaxsentan PK In Healthy Subjects
Brief Title: A Pharmacokinetic Drug-Drug Interaction (DDI) Study Between Sitaxsentan And Sildenafil, And Between Sitaxsentan And Tadalafil After Multiple Doses
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety Issue: The trial was prematurely terminated on Dec 9, 2010, due to safety concerns, specifically new emerging evidence of hepatic injury.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B1321056
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Results first posted 2012-02-22 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2011-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: A pharmacokinetic drug-drug interaction study between sitaxsentan and tadalafil and between sitaxsentan and sildenafil at the steady-state
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — sitaxsentan; Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): sitaxsentan 100 mg QD for 6 days (Treatment A)
  Interventions: Drug: sitaxentan
- Treatment B (Experimental): tadalafil 40 mg QD for 6 days
  Interventions: Drug: tadalafil
- Treatment C (Experimental): sitaxsentan 100 mg QD co-administered with tadalafil 40 mg QD for 6 days
  Interventions: Drug: sitaxsentan; Drug: tadalafil
- Treatment D (Experimental): sitaxsentan 100 mg QD co-administered with sildenafil 20 mg TID for 6 days
  Interventions: Drug: sitaxsentan; Drug: sildenafil

INTERVENTIONS:
Drug: sitaxentan — sitaxsentan 100 mg QD for 6 days
  Other Names: Thelin
  Arms: Treatment A
Drug: tadalafil — tadalafil 40 mg QD for 6 days
  Arms: Treatment B
Drug: sitaxsentan — sitaxsentan 100 mg QD for 6 days
  Arms: Treatment C
Drug: tadalafil — tadalafil 40 mg QD for 6 days
  Arms: Treatment C
Drug: sitaxsentan — sitaxentan 100 mg QD for 6 days
  Arms: Treatment D
Drug: sildenafil — sildenafil 20 mg TID for 6 days
  Arms: Treatment D

SUMMARY:
Sitaxsentan has a low drug-drug interaction potential and it did not have a clinically relevant effect on pharmacokinetics of sildenafil (a CYP3A sensitive substrate and PDE5 inhibitor).

Tadalafil did not have clinically relevant effect on pharmacokinetics of bosentan and ambrisentan. Based on overall clinical drug-drug interaction profiles, and in vitro CYP enzymes and transporter data, a clinically relevant drug-drug interaction between sitaxsentan and tadalafil is not expected. Sildenafil is not expected to affect sitaxsentan pharmacokinetics (PK), as sitaxsentan is a substrate of CYP3A4 and CYP2C9, where sildenafil did not show clinically relevant effect on PK of substrates of CYP3A4 and CYP2C9.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and women of non-child bearing potential between the ages of 21 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) or clinical findings at Screening.
* A positive urine drug screen.
* Subjects with hepatic dysfunction, defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >1.5 times the upper limit of the normal range at Screening. A retest may be done if AST and/or ALT within 1.5- to 2- times the upper limit of the normal range at Screening, and the average of the first and repeated test values should be used to decide the eligibility.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321056&StudyName=A%20Pharmacokinetic%20Drug-Drug%20Interaction%20%28DDI%29%20Study%20Between%20Sitaxsentan%20And%20Sildenafil%2C%20And%20Between%20Sitaxsentan%20And%20Tadalafil%20After%20Mult

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated for safety reasons (hepatoxicity) after dosing was completed for the first intervention.
Groups:
- Sitax, Then Tad, Then Sitax and Tad, Then Sitax and Sild: Sitaxsentan 100 milligram (mg) tablet once daily (QD) for 6 days, then tadalafil 40 mg tablet QD for 6 days, then sitaxsentan 100 mg tablet QD co-administered with tadalafil 40 mg tablet QD for 6 days, then sitaxsentan 100 mg tablet QD co-administered with sildenafil 20 mg table three times daily (TID) for 6 days. Only the first treatment in the sequence was administered due to the early termination.
- Tad, Then Sitax and Sild, Then Sitax, Then Sitax and Tad: Tadalafil 40 mg tablet QD for 6 days, then sitaxsentan 100 mg tablet QD co-administered with sildenafil 20 mg table TID for 6 days, then sitaxsentan 100 mg tablet QD for 6 days, then sitaxsentan 100 mg tablet QD co-administered with tadalafil 40 mg tablet QD for 6 days. Only the first treatment in the sequence was administered due to the early termination.
- Sitax and Tad, Then Sitax, Then Sitax and Sild, Then Tad: Sitaxsentan 100 mg tablet QD co-administered with tadalafil 40 mg tablet QD for 6 days, then sitaxsentan 100 mg tablet QD for 6 days, then sitaxsentan100 mg tablet QD co-administered with sildenafil 20 mg table TID for 6 days, then tadalafil 40 mg tablet QD for 6 days. Only the first treatment in the sequence was administered due to the early termination.
- Sitax and Sild, Then Sitax and Tad, Then Tad, Then Sitax: Sitaxsentan 100 mg tablet QD co-administered with sildenafil 20 mg table TID for 6 days, then sitaxsentan 100 mg tablet QD co-administered with tadalafil 40 mg tablet QD for 6 days, then tadalafil 40 mg tablet QD for 6 days, then sitaxsentan 100 mg tablet QD for 6 days. Only the first treatment in the sequence was administered due to the early termination.
Period: Overall Study
Arm/Group | Sitax, Then Tad, Then Sitax and Tad, Then Sitax and Sild | Tad, Then Sitax and Sild, Then Sitax, Then Sitax and Tad | Sitax and Tad, Then Sitax, Then Sitax and Sild, Then Tad | Sitax and Sild, Then Sitax and Tad, Then Tad, Then Sitax
Started | 4 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 4 | 4
Not completed — Study terminated | 4 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All randomized participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Median (Full Range); unit: hours
Groups:
- Sitaxsentan: Sitaxsentan 100 mg tablet QD for 6 days during any treatment period. Only the first treatment in the sequence was administered due to the early termination.
- Tadalafil: Tadalafil 40 mg tablet QD for 6 days during any treatment period. Only the first treatment in the sequence was administered due to the early termination.
- Sitaxsentan and Tadalafil: Sitaxsentan 100 mg tablet QD co-administered with tadalafil 40 mg tablet QD for 6 days during any treatment period. Only the first treatment in the sequence was administered due to the early termination.
- Sitaxsentan and Sildenafil: Sitaxsentan 100 mg tablet QD co-administered with sildenafil 20 mg tablet TID for 6 days during any treatment period. Only the first treatment in the sequence was administered due to the early termination.
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Trough Plasma Concentrations (Ctrough)
Description: Minimum or "trough"concentrations
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Geometric Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Geometric Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Area Under the Curve of the 24 Hour Dosing Interval (AUC24)
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Geometric Mean (Standard Deviation); unit: nanogram hour per milliliter (ng*hr/mL)
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Apparent Oral Clearance (CL/F)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Geometric Mean (Standard Deviation); unit: mL/minute
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Primary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Day 6 (predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose)
Population: Not analyzed due to early study termination.
Measure: Geometric Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another subject, or 1 participant may have experienced both a serious and nonserious event during the study.
Groups:
- Sitaxsentan: Sitaxsentan 100 mg tablet QD for 6 days
- Tadalafil: Tadalafil 40 mg tablet QD for 6 days
- Sitaxsentan and Tadalafil: Sitaxsentan 100 mg tablet QD co-administered with tadalafil 40 mg tablet QD for 6 days
- Sitaxsentan and Sildenafil: Sitaxsentan 100 mg tablet QD co-administered with sildenafil 20 mg table TID for 6 days
Arm/Group | Sitaxsentan | Tadalafil | Sitaxsentan and Tadalafil | Sitaxsentan and Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 4/4 | 4/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=4) | Tadalafil (N=4) | Sitaxsentan and Tadalafil (N=4) | Sitaxsentan and Sildenafil (N=4)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 3 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Study endpoints were not analyzed due to early termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.